CLINICAL TRIAL: NCT06074380
Title: Non Inferiority Trial Investigating Surfactants Administered Via MIST
Acronym: Niftisurf
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Matthew Derrick, Attending Neonatologist, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EH23-232
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: Pulmonary Surfactant; CPAP; Neonate
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Comparison of the efficacy of calfactant compared to poractant alfa administered with a minimally invasive method for the treatment of respiratory distress syndrome in 28-36 week infants
Who Masked: Participant, Investigator
Masking Description: Surfactant will be sent from Investigational Pharmacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calfactant (Infasurf) (Experimental): Neonate, 28-35 weeks gestation, less than 48 hours of age, with respiratory distress syndrome on CPAP > 30% oxygen will be given 3ml/kg of Calfacant
  Interventions: Drug: MIST surfactant
- Poractant alfa (Curosurf) (Experimental): Neonate, 28-35 weeks gestation, less than 48 hours of age, with respiratory distress syndrome on CPAP > 30% oxygen will be given 2.5ml/kg of Poractant alfa.
  Interventions: Drug: MIST surfactant

INTERVENTIONS:
Drug: MIST surfactant — Surfactant will be given via MIST while neonate is on CPAP

SUMMARY:
RESEARCH DESIGN Multicenter, randomized, controlled trial. RECRUITMENT Entry criteria Preterm infants 28-35 6/7 weeks' gestation and less than 48 hours of age who have a clinical diagnosis of respiratory distress syndrome. Infants who are on NCPAP and FiO2 ≥0.30 will randomized to curosurf or infasurf via MIST.

Exclusion criteria Infants will be excluded if there is a congenital anomaly or an alternative cause for respiratory distress.

Babies who require emergent intubation will not be enrolled in the interventions.

Parental Consent will be obtained prior to randomization.

DETAILED DESCRIPTION:
INTERVENTION Infants who on CPAP who reach the threshold of 30% oxygen will be randomized to calfactant (Infasurf), 3ml/kg or poractant alfa (Curosurf), 2.5ml/kg, administered under direct laryngoscopy using a surfactant instillation catheter (MIST) 16G Angiocath (Becton Dickinson, Sandy, UT, USA).

A second dose of calfactant (Infasurf) 3ml/kg or poractant alfa (Curosurf), 1.25ml/kg, will be administered via MIST their fiO2 reaches the threshold of 30% between 6 and 48 hours after the first dose.

No further surfactant should be given in the first 7 days unless the infant reaches the intubation criteria.

POST-INTERVENTION MANAGEMENT Other than the requirement to adhere to intubation criteria in the first week, and in some cases perform a room air trial at 36 weeks corrected gestation, management will be at the discretion of the clinical team.

Titration of CPAP pressure is encouraged, with a permitted maximum of 8 cm H2O. Use of nasal IPPV is allowable for apnea, but discouraged for RDS and should only be after at least one dose of surfactant has been given. Early caffeine therapy is expected.

Criteria for intubation:

Enrolled infants on CPAP will be intubated if:

* FiO2 ≥0.45 for 15 minutes, or if there is unremitting apnea (> 6 episodes/hour requiring intervention or in the opinion of the treating physician) or persistent respiratory acidosis (pH<7.25 and pCO2 >60) on blood gasses at least 30 minutes apart or metabolic acidosis refractory to treatment.
* Need for an anesthetic or an intervention requiring intubation

These criteria apply during the first week of life, and to the first episode of intubation only. If the infant is intubated it is expected that another dose of surfactant will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants 28-35 6/7 weeks' gestation and less than 48 hours of age who have a clinical diagnosis of respiratory distress syndrome confirmed by a chest x-ray on nasal continuous positive airway pressure (NCPAP) and FiO2 ≥0.30

Exclusion Criteria:

* Infants will be excluded if there is a congenital anomaly or an alternative cause for respiratory distress.
* Infants who require emergent intubation will not be enrolled in the interventions.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 262 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of infants requiring Endotracheal Intubation | 7 days
  Infants will have an endotracheal placed if their inspired oxygen is >45% for more than 15 minutes

SECONDARY OUTCOMES:
Duration of positive pressure support | 36 weeks corrected gestational age
  Endotracheal ventilation or Non-invasive Ventilation or CPAP or NC flow>2 L
Duration of Supplemental oxygen | 36 weeks corrected gestational age
  Oxygen requirement to keep saturations >95%

CONTACTS AND LOCATIONS:
Locations (1):
- Northshore University Healthsystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dargaville PA, Kamlin COF, Orsini F, Wang X, De Paoli AG, Kanmaz Kutman HG, Cetinkaya M, Kornhauser-Cerar L, Derrick M, Ozkan H, Hulzebos CV, Schmolzer GM, Aiyappan A, Lemyre B, Kuo S, Rajadurai VS, O'Shea J, Biniwale M, Ramanathan R, Kushnir A, Bader D, Thomas MR, Chakraborty M, Buksh MJ, Bhatia R, Sullivan CL, Shinwell ES, Dyson A, Barker DP, Kugelman A, Donovan TJ, Tauscher MK, Murthy V, Ali SKM, Yossuck P, Clark HW, Soll RF, Carlin JB, Davis PG; OPTIMIST-A Trial Investigators. Effect of Minimally Invasive Surfactant Therapy vs Sham Treatment on Death or Bronchopulmonary Dysplasia in Preterm Infants With Respiratory Distress Syndrome: The OPTIMIST-A Randomized Clinical Trial. JAMA. 2021 Dec 28;326(24):2478-2487. doi: 10.1001/jama.2021.21892. PMID 34902013
- [Background] Kribs A, Hartel C, Kattner E, Vochem M, Kuster H, Moller J, Muller D, Segerer H, Wieg C, Gebauer C, Nikischin W, Wense Av, Herting E, Roth B, Gopel W. Surfactant without intubation in preterm infants with respiratory distress: first multi-center data. Klin Padiatr. 2010 Jan-Feb;222(1):13-7. doi: 10.1055/s-0029-1241867. Epub 2010 Jan 18. PMID 20084586